CLINICAL TRIAL: NCT05993000
Title: Effect Of Mobilization, Exercise And Music On Frozen Shoulder Patients
Brief Title: Assessment of Frozen Shoulder Treatment Using 432 Hertz Frequency Music: A Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, SELMA İŞLER, Physiotherapist, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NEHIR55
Record Dates: First submitted 2023-07-30; First posted 2023-08-15 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Frozen Shoulder; 432 Hertz Frequency Music; Manual Therapy; Exercise
Keywords: Frozen Shoulder; 432 Hertz Frequency Music; Manual Therapy
MeSH Terms: conditions — Bursitis; Motor Activity | interventions — Transcutaneous Electric Nerve Stimulation; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Grup 1(Music + mobilization + exercise was applied) (Experimental): In this group, hot packs and TENS (Transcutaneous Electrical Nerve Stimulation) were applied to the patients simultaneously, while they were listening to 432 hertz frequency music through headphones. Subsequently, shoulder mobilization was applied in appropriate positions. The exercises were conducted by the physiotherapist during the session and the manageable exercises were given to the patients as a home program.
  Interventions: Other: 432 Hertz frequency music; Other: TENS; Other: Mobilization; Other: Exercises; Other: Hotpack
- Grup 2 ( music + exercise) (Experimental): In this group, hot packs and TENS (Transcutaneous Electrical Nerve Stimulation) were applied to the patients simultaneously, while they were listening to 432 hertz frequency music through headphones. The exercises were conducted by the physiotherapist during the session and the manageable exercises were given to the patients as a home program.
  Interventions: Other: 432 Hertz frequency music; Other: TENS; Other: Exercises; Other: Hotpack
- Grup 3 (mobilization + exercise) (Active Comparator): After applying hot packs and TENS(Transcutaneous Electrical Nerve Stimulation) to the patients, shoulder mobilization was performed in suitable positions.The exercises were conducted by the physiotherapist during the session and the manageable exercises were given to the patients as a home program.
  Interventions: Other: TENS; Other: Mobilization; Other: Exercises; Other: Hotpack
- Grup 4 (exercise) (Active Comparator): After the application of hot packs and TENS (Transcutaneous Electrical Nerve Stimulation) to the patients, the physiotherapist administered specific exercises during the session. Additionally, customized exercises were prescribed as a home program for the patients to continue their rehabilitation outside of the clinic setting.
  Interventions: Other: TENS; Other: Exercises; Other: Hotpack

INTERVENTIONS:
Other: 432 Hertz frequency music — 432 Hertz frequency music was played to patients through headphones during hotpack and TENS applications.
  Arms: Grup 1(Music + mobilization + exercise was applied); Grup 2 ( music + exercise)
Other: TENS — The TENS treatment was conducted using a double-channel TENS device equipped with four electrodes. The electrodes were placed around the painful area to ensure targeted stimulation. Each session lasted for 30 minutes, during which the TENS device operated at a high frequency range of 60-120 Hz. To achieve the desired analgesic effect, a short transition time of 20-120 microseconds was employed.
Other: Mobilization — Electrophysiological agents were administered to the affected shoulder joint area before initiating mobilization. The Cyriax mobilization techniques targeted the scapula, clavicular, and GH joints, considering their biomechanical interaction and the specific dysfunction of each patient.
  Arms: Grup 1(Music + mobilization + exercise was applied); Grup 3 (mobilization + exercise)
Other: Exercises — The combined utilization of exercises targeting the glenohumeral (GH) joint, scapulothoracic (ST) region, and stretching has demonstrated significant effectiveness in ameliorating range of motion and alleviating pain during the treatment of Frozen Shoulder (FS). These exercises were closely supervised and administered by the physiotherapist in each session. Furthermore, a home exercise program was provided to the patients, consisting of exercises for posture, thera band, and finger ladder. They were instructed to perform 10-15 repetitions of these exercises twice a day independently.
Other: Hotpack — Each group of patients received a 20-minute hot pack application to the scapula and shoulder circumference.

SUMMARY:
The goal of this clinical trial is to determine the effect of listening to music during the treatment of frozen shoulder on pain, normal range of motion, functional activity status and quality of life.Upon recruitment, the subjects were randomly assigned to one of four treatment groups: Group 1 received Music + Mobilization + Exercise, Group 2 received Music + Exercise, Group 3 received Mobilization + Exercise, and Group 4 received Exercise only.

DETAILED DESCRIPTION:
Forty individuals diagnosed with frozen shoulder were randomly allocated into four distinct treatment groups. Each participant received a total of eighteen treatment sessions, administered three days per week. Pain levels, range of motion of the shoulder joint, functional status, general health condition, and quality of life were measured and recorded for each participant both before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic or primary adhesive capsulitis5,20,32,
* a diagnosis of stage 2-3,
* unilateral condition,
* age between 30 to 65 years,
* normal findings on radiographs within the previous 12 months,
* no previous shoulder surgeries to the affected shoulder,
* no previous manipulations under anesthesia of the affected shoulder,
* passive joint movements limited to 50-75% of the normal range of motion of the joint, - and no hearing loss.

Exclusion Criteria:

* have shoulder girdle motor control deficits associated with neurological disorders.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-05-29 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Goniometer | baseline and 6 weeks
  A goniometer was used to measure the participants' shoulder range of motion.
Visual Analog Scale | baseline and 6 weeks
  The Visual Analog Scale is a psychometric response scale used to measure subjective characteristics or attitudes, and it has been utilized to assess the pain levels of participants.10-cm visual analog scale, ranging from 0 ("no pain") to 10 ("the worst imaginable pain").
Disabilities of the Arm, Shoulder, and Hand | baseline and 6 weeks
  I used this scale to evaluate the participants' upper extremity functions.The questionnaire consists of 30 items that cover various activities related to daily living, work, and recreational activities that involve the use of the upper extremities. Participants rate their ability to perform each activity and the severity of their symptoms on a scale from 1 to 5, where 1 represents "no difficulty" or "no symptoms" and 5 represents "unable to do" or "extremely severe symptoms."A high score means that the patient's condition is poor.
Modified Constant Score | baseline and 6 weeks
  The questionnaire used to measure muscle strength was applied because the participants had shoulder joint range of motion less than 90 degrees before treatment.The Modified Constant Score typically evaluates four main components:
  Pain ( 0 being no pain and 15 being severe pain),Activities of Daily Living (20 points: This section assesses the patient's ability to perform various activities using the affected shoulder, such as combing hair, putting on a coat, and reaching behind the back), Strength ( The examiner rates the strength on a scale from 0 to 25), Range of Motion (40 points). The total Modified Constant Score is the sum of the points obtained in each of these four components, resulting in a maximum score of 100. Higher scores indicate better shoulder function and range of motion.
36-Item Short Form Health Survey | baseline and 6 weeks
  Anket used to assess the overall health status of the participants is the "36-Item Short Form Health Survey" or "SF-36.The SF-36 consists of 36 questions that cover eight health domains:
  Physical Functioning, Role Limitations due to Physical Health Problems,Bodily Pain,General Health,Vitality, Social Functioning,Role Limitations due to Emotional Problems, Mental Health.
  Each domain is assessed through multiple questions, and the responses are scored and transformed to create summary scores for each domain. These summary scores can range from 0 to 100, with higher scores indicating better health-related quality of life.

SECONDARY OUTCOMES:
BMI(Basal Mass Index) | baseline and 6 weeks
  BMI is a measure that assesses the relationship between a participants weight and height. BMI is calculated using weight in kilograms and height in meters.
  The formula for calculating BMI is as follows:
  BMI = Weight (kg) / (Height)^2 (m^2)

CONTACTS AND LOCATIONS:
Overall Officials: SELMA İŞLER, Phd, Principal Investigator — Ondokuz Mayıs University; Seydi Ahmet Ağaoğlu, Prof., Study Director — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayıs University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 2 years
Access Criteria: Researchers at universities